CLINICAL TRIAL: NCT02533518
Title: Ultra-Violet Fluorescence Bronchial Cancer Location
Acronym: UVFBCL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1008041; 2010-A00343-36 (Other: AFSSAPS)
Record Dates: First submitted 2015-08-17; First posted 2015-08-26 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients with lung cancer (Experimental)
  Interventions: Procedure: Rigid bronchoscopy with ultraviolet transmission; Other: Biopsy

INTERVENTIONS:
Procedure: Rigid bronchoscopy with ultraviolet transmission
Other: Biopsy

SUMMARY:
Diagnose lung cancer at an early stage is crucial for effective treatment. At these early stages, cancer is usually invisible in ambient white light when the endoscopic analysis of the bronchial mucosa. This lining is self-fluorescent at its illumination by blue light. These widely distributed autofluorescence methods detect early mucosal abnormalities. They are very sensitive but not specific to recognize the lung cancer. Thanks to European funding (EURIMUS), a new tool with fluorescent UV light has been developed.

The purpose of this preliminary study is to verify the suitability for specific detection of cancerous tissue in Pneumology of this fluorescence method versus histological analysis of the tissue.

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated or entitled to a social security scheme
* Major Patient
* Patient who signed the informed consent document
* Patient with a known primary cancer in bronchial level

Exclusion Criteria:

* Pregnant woman
* Patient with a benign tumor histology
* Patient with an unknown tumor histology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
ultraviolet fluorescence ratio Iodine360 / Iodine450 | Day 0
  Detection of cancerous tissues and healthy or inflammatory tissues is used to calculate the sensitivity and specificity of the rigid bronchoscopy with UV transmission compared to biopsy (gold standard).
Histology of tissue | Day 0
  The histology give the final diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Pneumology departement CHU Saint-Etienne, Saint-Etienne, France